CLINICAL TRIAL: NCT06042842
Title: The Value of circRNAs (hsa_circ_0004001) in Early Diagnosis of HCC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Aboelim Shafeik, msc of clinical batology, Assiut University
Other Study IDs: CircRNA in HCC
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Hepatic Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- group 1: healthy control
- group 2: patient with hepatic cell carcinoma
- group 3: patient with non malignant liver diseased

SUMMARY:
1. To evaluate the clinical utility of plasma circRNAs (hsa_circ_0004001) as a non invasive diagnostic biomarker for HCC patients and to differentiate between malignant and nonmalignant hepatic disorders.
2. To study the relation of circRNAs (hsa_circ_0004001) to HCC staging.
3. To compare between circRNAs (hsa_circ_0004001) and the routine marker (AFP) as biomarkers for HCC diagnosis.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the most common malignant gastrointestinal tumours worldwide and is characterized by high morbidity and mortality rates . HCC is the sixth common cancer and the second leading cause of death from cancer worldwide.

The American Cancer Society's estimates for deaths by primary liver cancer and intrahepatic bile duct cancer in the United States for 2018 are 30200. HCC incidence in Egypt has increased sharply over the last decade due to the high prevalence of hepatitis B virus (HBV) and hepatitis C virus (HCV) infection among Egyptians. Indeed, liver cancer is the most frequent cancer in both men and women in Egypt. HCC was the first among the most frequently observed cancers in lower and middle Egypt and the 2nd in upper Egypt, of patients with liver cirrhosis, 3%-5% develop HCC annually. In Egypt, HCC represents nearly 70% of all liver tumors.

Unfortunately, upon diagnosis, most of the patients are in the advanced stages of the disease. Thus, early diagnosis is a key in improving the HCC treatment and prognosis. Liver cancer screening is typically based on the detection of serum alpha-fetoprotein and various imaging methods. Moreover, imaging techniques are costly, and the patients' compliance is poor. The diagnostic and treatment strategies that are available for HCC, it still cannot be detected at early stages efficiently. The diagnostic methods fail to detect HCC in many patients. Consequently, curative treatments may no longer be efficient at the time of diagnosis because of intra- and extrahepatic metastases. The combination of serum alpha-fetoprotein (AFP) and ultrasound surveillance is the most widely used method for screening and detection of HCC in high-risk groups. However, ultrasound surveillance is limited by the sensitivity of the detection and often results in misdiagnosis of small malignant nodules, especially in cirrhosis. Therefore, due to their poor sensitivity and specificity, there is a great need to improve the current HCC diagnostic methods. The search for novel potential biomarkers is crucial to increase the rate of early detection.

Circular RNAs (circRNAs) are a type of single-stranded RNA which, unlike linear RNA, forms a covalently closed continuous loop. In circular RNA, the 3' and 5' ends normally present in an RNA molecule have been joined together. Because circular RNA does not have 5' or 3' ends, it is resistant to exonuclease-mediated degradation and is presumably more stable than most linear RNA in cells. They are covalently closed loops generated by the back splicing of precursor mRNA (premRNA) molecules, which exist widely in mammalian cells and are characterized by stability, conservative evolution, and cell or tissue specificity. These characteristics endow circRNAs with many biological functions, such as acting as microRNA (miRNA) sponges, regulating the transcription of parental genes, binding RNA binding proteins (RBPs), and encoding proteins and peptides. The circRNA is a type of non-coding RNA and type of nucleic acid molecule found in exosomes, forms a covalently bonded closed loop without 5' caps or 3' poly(A) tails. Most circRNAs have the following characteristics: (1) High abundance: The abundance of circRNA expression varies greatly; in some cases, the abundance of circRNAs exceeds 10 times that of their linear RNA counterparts; (2) Stability: The stability of circRNAs is 2.5-5 times higher than that of linear transcripts because the unique covalently closed loop of circRNAs lacks 3' and 5' ends, resulting in the absence of ribonuclease binding targets; therefore, circRNAs are not easily degraded; (3) Conservation: CircRNAs are widely present in different species and are evolutionarily conserved. Some studies suggest that most circRNAs in different species are evolutionarily conserved, while a few are not conserved ; and (4) Specificity: CircRNAs have tissue and cell specificity, with differential expression in different stages of ontogeny and disease progression .

They are superior to other non-coding RNAs as molecular diagnostic markers and drug treatment targets. Exosomal-derived circRNAs in the body fluids of tumours patients can modulate tumour proliferation, invasion, metastasis, and drug resistance. They can be used as effective biomarkers for early non-invasive diagnosis and prognostic evaluation of tumours and represent ideal targets for early precision therapeutic intervention. The circRNA secreted into human circulating blood can be used as a biomarker for disease diagnosis . Our knowledge of the pathogenesis of hepatocellular carcinoma (HCC) is incomplete. The effective treatment methods are surgery or transplantation, but the recurrence and metastasis rates are still high with a low 5-year survival rate . Many circRNAs are involved in the proliferation, apoptosis, migration, and invasion of HCC cells. Therefore, circRNA may be an important biomarker for the clinical diagnosis and treatment of HCC. According to the effect on the malignant phenotype of HCC cells, circRNAs can be divided into carcinogenic circRNAs and tumor suppressor circRNAs. Compared with the adjacent tissues and normal liver cell lines, the expression of cancer-promoting circRNAs in HCC tissues and HCC cell lines is usually high. Inhibiting the expression of carcinogenic circRNAs can significantly reduce the proliferation, migration, and invasion of HCC cells, promote the apoptosis of HCC cells, and improve the prognosis Recent studies demonstrated that numerous circRNAs were differentially expressed in HCC tissues, which is closely related with the development and prognosis of HCC, and indicated that circRNA plays vital roles in tumorigenesis and progression of HCC and could be used as a diagnostic biomarker

ELIGIBILITY:
Inclusion Criteria:

1. group one patients early diagnosed as HCC
2. group two patient diagnosed with chronic non-malignant liver disease 3 group three healthy control group

Exclusion Criteria:

1. Patients with any other type of malignant or benign tumors should be excluded from our study.
2. History of chemotherapy or surgical treatment of cancer

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: (102 )individuals aged (18 years to 80years), did not receive any chemotherapy or surgical treatment The study will be carried out on patients who will be admitted to gastroenterology department at Assiut University hospital, and will be conducted at clinical pathology department, Assiut University Hospital, Faculty of medicine, Assiut University
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
(1) To evaluate the clinical utility of plasma circRNAs (hsa_circ_0004001)by Q-PCR as a non invasive diagnostic biomarker for HCC patients and to differentiate between malignant and nonmalignant hepatic disorders | baseline
  1. To evaluate the clinical utility of plasma circRNAs (hsa_circ_0004001) by Q-PCR as a non invasive diagnostic biomarker for HCC patients and to differentiate between malignant and nonmalignant hepatic disorders
  2. To study the relation of circRNAs (hsa_circ_0004001) to HCC staging.
  3. To compare between circRNAs (hsa_circ_0004001) and the routine marker (AFP) as biomarkers for HCC diagnosis